CLINICAL TRIAL: NCT02743091
Title: Idiopathic Pre-capillary Pulmonary Hypertension in Patients With End-stage Kidney Disease
Brief Title: Idiopathic Pre-capillary Pulmonary Hypertension in ESKD Patients
Status: Completed | Type: Observational
Sponsor: Toujinkai Hospital (Other)
Responsible Party: Principal Investigator, Masato Nishimura, MD, Director of Cardiovascular Division, Toujinkai Hospital
Other Study IDs: PHdialysis
Record Dates: First submitted 2016-04-06; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Hypertension
Keywords: heart failure; survival; end-stage kidney disease
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study investigates the prevalence and prognosis of idiopathic pre-capillary pulmonary hypertension (PH) in patients with end-stage kidney disease (ESKD).

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a rare cardiovascular disease with progressive and fatal features. PH is classified into the 5 groups, and the prevalence of group 1 pulmonary arterial hypertension, including idiopathic and heritable, is 5 to 15 cases per one million adults and a median survival was reportedly three years. PH found in patients with end-stage kidney disease (ESKD) is classified into group 5, because the pathogenesis and clinical characteristics have not been clarified. The prevalence of PH in patients with ESKD was reportedly around 17~56% based on echocardiographic studies. In this study, we evaluated the incidence of idiopathic pre-capillary PH of ESKD patients by right heart catheterization, and examined the prognosis by following the occurrence of heart failure death.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of dyspnea, hypotension (systolic blood pressure <90mmHg, or syncope.
* Systolic pressure gradients in tricuspid valve of 40 mmHg or more.
* In right heart catheterization, precapillary PH was defined as mean pulmonary arterial pressure (PAP) ≥25 mmHg, pulmonary vascular resistance (PVR) ≥3 wood unit, and pulmonary artery wedge pressure (PAWP) ≤15 mmHg.

Exclusion Criteria:

* Patients with systolic left ventricular dysfunction (left ventricular ejection fraction [LVEF] <50%), mitral or aortic regurgitation of grade 2 or more, aortic or mitral surface <1.5 cm2, severe anemia (blood hemoglobin <9 g/dl), severe chronic obstructive pulmonary disease defined by percent predicted forced expiratory volume in one second <60%, or lung fibrosis were not enrolled in this study.
* In right hear catheterization, PAP ≥25 mmHg and PAWP >15 mmHg were diagnosed as post capillary PH.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ESKD who had received medical treatment at pre-dialysis stage or had undergone maintenance hemodialysis in Toujinkai Hospital from January 1, 2001 to December 31, 2014
Sampling Method: Non-Probability Sample
Enrollment: 1988 (Actual)
Dates: Start 2001-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients of idiopathic pre-capillary hypertension | 14 years

SECONDARY OUTCOMES:
Number of patients who died of heart failure | 14 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nishimura M, Tokoro T, Yamazaki S, Hashimoto T, Kobayashi H, Ono T. Idiopathic pre-capillary pulmonary hypertension in patients with end-stage kidney disease: effect of endothelin receptor antagonists. Clin Exp Nephrol. 2017 Dec;21(6):1088-1096. doi: 10.1007/s10157-016-1344-y. Epub 2016 Oct 19. PMID 27757709